CLINICAL TRIAL: NCT04336839
Title: Vascular Resection During Pancreaticoduodenectomy for Pancreatic Neuroendocrine Neoplasms (PanNENs): a Comparative Single Centre Study
Brief Title: Portal Vein Resection in Pancreatic Neuroendocrine Tumours
Acronym: PVNET
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 11536
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Pancreas Neoplasm; Neuroendocrine Tumors
Keywords: portal vein resection; pancreatic surgery
MeSH Terms: conditions — Pancreatic Neoplasms; Neuroendocrine Tumors | interventions — Plastic Surgery Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Portal vein resection / reconstruction — Portal vein resection and reconstruction, with or without concommitant arterial resection

SUMMARY:
The limited evidence on the value of portal vein resection in patients with borderline resectable and/or locally advanced PanNENs is an incentive to carry out a retrospective multicentre study amongst centres with specific interest in the management of PanNENs and with experience on vascular reconstruction. Unlike previous studies on pancreatic cancer, it is more difficult to standardise the comparative parameters as the definition of borderline resectable disease has never been published for PanNENs. Similarly, different histological classifications make impossible to collect data exclusively on T3 tumours. Therefore, we aim to compare the short and long-term outcomes (including the impact of the histological depth of vascular invasion on survival) between patients undergoing standard PD and PD with portal vein resection for PanNENs, (regardless of T stage), by collecting and analysing retrospective data in this single centre study

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing pancreaticoduodenectomy (Whipple's or Pylorus Preserving Pancreaticoduodenectomy) for sporadic PanNENs of the head of the pancreas of any stage (R0 or R1 resections) operated from 1st January 2007 up to 31st December 2016 inclusive.

Exclusion Criteria:

* Multiple Neuroendocrine Neoplasia (MEN) syndrome or other genetic background
* Age <18 years old
* Total pancreatectomy or different operation rather than PD
* R2 Resections

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients operated for pancreatic neuroendocrine tumours within a single tertiary referal centre
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | total of 2 years retrospective follow up
  Time from surgery to disease progression, or death or completion of follow up

SECONDARY OUTCOMES:
Morbidity and mortality rate | total of 2 years retrospective follow up
  Postoperative morbidity and mortality
Histology predictive value | total of 2 years retrospective follow up
  Predictive value of histologically proven invasion of the portal vein adventitia

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe K Fusai, MD MS, Principal Investigator — Royal Free London NHS Foundation Trust & University College London

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers

REFERENCES:
- [Result] Sakamoto E, Hasegawa H, Ogiso S, Igami T, Mori T, Mizuno T, Hattori K, Sugimoto M, Fukami Y. Curative resection for a pancreatic endocrine carcinoma involving the portal vein. Hepatogastroenterology. 2004 Nov-Dec;51(60):1849-51. PMID 15532841
- [Result] Touzios JG, Kiely JM, Pitt SC, Rilling WS, Quebbeman EJ, Wilson SD, Pitt HA. Neuroendocrine hepatic metastases: does aggressive management improve survival? Ann Surg. 2005 May;241(5):776-83; discussion 783-5. doi: 10.1097/01.sla.0000161981.58631.ab. PMID 15849513
- [Result] van Geenen RC, ten Kate FJ, de Wit LT, van Gulik TM, Obertop H, Gouma DJ. Segmental resection and wedge excision of the portal or superior mesenteric vein during pancreatoduodenectomy. Surgery. 2001 Feb;129(2):158-63. doi: 10.1067/msy.2001.110221. PMID 11174708
- [Result] Ravikumar R, Sabin C, Abu Hilal M, Bramhall S, White S, Wigmore S, Imber CJ, Fusai G; UK Vascular Resection in Pancreatic Cancer Study Group. Portal vein resection in borderline resectable pancreatic cancer: a United Kingdom multicenter study. J Am Coll Surg. 2014 Mar;218(3):401-11. doi: 10.1016/j.jamcollsurg.2013.11.017. Epub 2013 Nov 27. PMID 24484730
- [Result] Elberm H, Ravikumar R, Sabin C, Abu Hilal M, Al-Hilli A, Aroori S, Bond-Smith G, Bramhall S, Coldham C, Hammond J, Hutchins R, Imber C, Preziosi G, Saleh A, Silva M, Simpson J, Spoletini G, Stell D, Terrace J, White S, Wigmore S, Fusai G. Outcome after pancreaticoduodenectomy for T3 adenocarcinoma: A multivariable analysis from the UK Vascular Resection for Pancreatic Cancer Study Group. Eur J Surg Oncol. 2015 Nov;41(11):1500-7. doi: 10.1016/j.ejso.2015.08.158. Epub 2015 Aug 28. PMID 26346183